CLINICAL TRIAL: NCT04263064
Title: Effect of Clonidine on High Volume-Low Concentration Caudals
Brief Title: High Volume Caudal Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Christopher Heine, MD, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00091670
Record Dates: First submitted 2020-02-01; First posted 2020-02-10 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Male Circumcision
MeSH Terms: interventions — Clonidine

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, observer blinded study will attempt to determine if there is any benefit to the addition of clonidine to a HVLC caudal block, both in duration of analgesia and occurrence of emergence agitation.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessor and patient blinded to the medications in the block that the patient receives.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High Volume-Low Concentration without Clonidine (Active Comparator): The control for this study will be a High Volume-Low Concentration (1.5cc/kg of 0.15% ropivacaine and 5mcg/cc epinephrine).
  Interventions: Drug: High Volume-Low Concentration without Clonidine
- High Volume-Low Concentration with clonidine (Experimental): The study intervention will be High Volume-Low Concentration with clonidine (1.5cc/kg of 0.15% ropivacaine, with 1mcg/cc of clonidine and 5mcg/cc epinephrine).
  Interventions: Drug: High Volume-Low Concentration with clonidine

INTERVENTIONS:
Drug: High Volume-Low Concentration without Clonidine — The control for this study will be a High Volume-Low Concentration (1.5cc/kg of 0.15% ropivacaine and 5mcg/cc epinephrine) caudal block
  Arms: High Volume-Low Concentration without Clonidine
Drug: High Volume-Low Concentration with clonidine — The study intervention will be High Volume-Low Concentration with clonidine (1.5cc/kg of 0.15% ropivacaine, with 1mcg/cc of clonidine and 5mcg/cc epinephrine).
  Arms: High Volume-Low Concentration with clonidine

SUMMARY:
The primary objective is to evaluate the effect of clonidine on the duration of analgesia provided by a high volume-low concentration caudal block for pediatric aurgical procedres. In addition, caudal clonidine's effect on length of recovery and post-operative emergence agitation will be measured.

ELIGIBILITY:
Inclusion Criteria:

* 3 years old or less
* Weight <= 13.3kg
* American Society of Anesthesiology Physical Status (ASA) 1 or 2
* Undergoing circumcision surgery
* Patients whose plan of care includes caudal block

Exclusion Criteria:

* Known allergy to clonidine, epinephrine, or amide local anesthetics
* Inability or unwillingness of parent or legal guardian to give informed consent

Ages: 0 Years to 3 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — presenting for penile circumcision
Enrollment: 129 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Presence of Pain | 24 hours
  The effect of clonidine on the duration of the analgesia provided by a high volume-low concentration caudal will be measured in the Post Anesthesia Care Unit pain assessments using CHEOPS score every at 0, 30, 60, and 90 minutes after arrival to PACU.
  The CHEOPS pain score tool is an observational scale for measuring postoperative pain in children aged 1-7 yrs. The tool includes six categories of pain behavior, each with 3-4 levels and scores range from 4 points (no pain) to 13 points (the worst pain).
Administration of Rescue Pain Medications | 24 hours
  Data will be collected and analyzed on the need for rescue pain medications by collecting doses of opioids administered the Post Anesthesia Care Unit.
Time to first Administration of Acetaminophen | 24 hours
  24 hours after discharge a phone call interview will be conducted to obtain the time of the first dose of acetaminophen

SECONDARY OUTCOMES:
Hemodynamic Changes | 24 hours
  A change of greater than 20% in heart rate or blood pressure from their baseline established in the preoperative area
Incidence of Emergence Delirium | 24 hours
  The incidence of emergence delirium will be collected utilizing the PAED Scale at 0, 30, 60, and 90 minutes after arrival to the Post Anesthesia Care Unit. The PAED scale will measure the presence of delirium by scoring behaviors from 1-4 (1=calm, 2=not calm but consolable, 3=moderately agitate, restless or not easily calmed, 4=combative, excited, thrashing around)
Sedation Levels | 24 hours
  Measured in PACU utilizing Ramsay Sedation Scale at 0, 30, 60, and 90 minutes after arrival in PACU. The Ramsay sedation scale is a scoring of responses (1-6) [1=anxious or restless, 2=cooperative, oriented, tranquil, 3=responding to commands, 4=brisk response to stimulus, 5=sluggish response to stimulus, 6=no response to stimulus].
Average Time to Discharge | 24 hours
  time of arrival to PACU and discharge time

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Heine, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No